CLINICAL TRIAL: NCT03659864
Title: The Role of Eicosanoids in the Cardiovascular Actions of Inhaled Nanoparticles
Acronym: ECOARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AC18026; SP/15/8/31575 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2018-08-09; First posted 2018-09-06 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Blood Biomarkers; Vasodilation; Blood Clotting; Lung Function; Healthy Volunteers
Keywords: nanoparticles; pollution
MeSH Terms: conditions — Aneurysm; Thrombosis | interventions — 1-(2-(dodecyloxy)ethyl)pyrrolidine hydrochloride; Soot

STUDY DESIGN:
Intervention Model Description: Cohort study with double blind randomised cross over design
Who Masked: Participant, Investigator
Masking Description: Participant and lead clinical fellow will be blinded. All staff involved in initial data generation will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure 1 (Sham Comparator): filtered air
  Interventions: Other: filtered air
- Exposure 2 (Experimental): nanoparticle 1 (either DEP or s-GO depending on group)
  Interventions: Other: diesel exhaust particulate; Other: small graphene oxide
- Exposure 3 (Experimental): nanoparticle 2 (either CB or us-GO depending on group)
  Interventions: Other: carbon nanoparticles; Other: ultrasmall graphene oxide

INTERVENTIONS:
Other: diesel exhaust particulate — aerosolised diesel exhaust particulate
  Other Names: DEP; SRM2975
  Arms: Exposure 2
Other: carbon nanoparticles — aerosolised 'clean' carbon nanoparticles
  Other Names: carbon black; CB; Printex 90
  Arms: Exposure 3
Other: small graphene oxide — aerosolised 'small' graphene oxide
  Other Names: s-GO
  Arms: Exposure 2
Other: ultrasmall graphene oxide — aerosolised 'ultrasmall' graphene oxide
  Other Names: us-GO
  Arms: Exposure 3
Other: filtered air — control: filtered air
  Other Names: FA
  Arms: Exposure 1

SUMMARY:
Nanoparticles (NPs) are minute pieces of material to which we are exposed every day in the air we breathe. Some are naturally occurring and have no impact on health, whereas others are produced from urban air pollution and can worsen diseases, particularly in the lungs and blood vessels. However, there is great interest in developing new NPs because of their unique properties that are useful for many applications, such as engineering, electronics and for drug delivery. At present it is unclear exactly what effects inhaled NPs have. Our current programme of research is designed to assess whether a specialized group of fats made in the body (called eicosanoids) drive the cardiovascular effects of NPs. The changes in the profiles of these fats will provide unique fingerprints that could be used to predict the actions of new NPs.

In the proposed clinical study we shall investigate the effects of both environmental and manufactured carbonaceous NPs on the lungs, blood vessels, blood clotting, and levels of eicosanoids in blood and urine. We have previously investigated the cardiovascular effects of carbon nanoparticles after inhalation in man, and these experiments will investigate how the shape, size and composition of carbon particles influence these responses. These experiments will provide new insight into how NPs affect the body and pave the way for new ways to predict the toxic effects of NPs (reducing the need for animal experiments). The findings will enable the design of novel NP without the harmful characteristics of those found in air pollution.

DETAILED DESCRIPTION:
This study will investigate the biological effects of inhaling different nanoparticles in healthy volunteers. We will compare 4 different types of nanoparticles: diesel exhaust nanoparticles (a nanoparticle with a complex mixture of chemicals), carbon black nanoparticles (a 'simple, clean' carbon nanoparticle) and two different sizes of graphene oxide (flat flakes of carbon), as well as inhalation of filtered air for comparison. Volunteers will be split randomly into 2 groups and each will be exposed to 3 nanoparticles, separately in a randomised order, with at least 2 weeks between the exposures (Cohort study with double blind randomised cross over design).

Screening visit 30 healthy non-smoking volunteers will be recruited. The volunteer will attend a screening visit at the Clinical Research Facility (CRF) at the Royal Infirmary of Edinburgh (RIE). Eligibility will be confirmed and consent taken. Baseline measurements of lung function (FEV1, FVC), blood pressure and blood biochemistry will be made. The participant will be asked to perform a short exercise test on a stationary bicycle to determine the bicycle workload for the main study.

Study visit On each visit, baseline measures will be taken at the CRF. The participant will be taken to a mobile facility to breathe in a set level of nanoparticles (target concentration of 200 micrograms per cubic metre) via a facemask for 2 hours while intermittently cycling. The mobile exposure chamber allows for volunteers to inhale specific air pollutants (typical of an urban environment), nanoparticles or gases at precise concentrations while exercising. Nanoparticles will be obtained as standard reference materials or by custom synthesis at the National Graphene Institute at the University of Manchester. All suspensions of nanoparticles are well characterised, free of contamination and have been extensively tested in preclinical models.

After the exposure the participant will return to the CRF and lung function and blood pressure re-measured. Blood will be withdrawn through a cannula in a large vein in the arm at set times after the exposure (15 min, 2h, 4h) for measurement of eicosanoids and other indicators of a haematological response (e.g. an inflammatory response). Blood will be slowly withdrawn (10 mL/min for 5 min) through a tube into a small piece of equipment called a Badimon Chamber which gives a measure of how readily the blood clots. The responsiveness of blood vessels in the arm will then be measured by a technique called forearm plethysmography. Here cuffs are inflated around the wrist and top of the arm and the blood flow is measured by a sensitive gauge around the forearm. Two different vasodilator drugs (acetylcholine and sodium nitroprusside) will be infused into an artery in the arm to see how the nanoparticle exposure has altered the way the blood vessels of the arm respond to these drugs. Blood will also be taken after each drug to measure substances that are release from the wall of arteries to give further indication of the health of the artery. The cannula will be removed and lung function and blood pressure will be re-measured. The participant will be allowed to rest, provided with food and drink, before leaving the hospital.

Biological samples (blood and urine) will be used to measure a range of cardiovascular parameters at the RIE and the University of Edinburgh. The primary endpoint for the study is the measurement of a panel of lipid mediators called eicosanoids, which will be performed by our collaborators at the University of Highlands and Islands who have specialised lipidomic facilities and experience in this area.

Shortened protocol An additional 12 volunteers will be recruited to perform a shortened version of the main protocol. The protocol is identical to the above with the exception that the forearm blood flow, Badimon study and the t=4 time point have been removed. These studies will be used to allow additional monitoring of the effect of nanoparticles during initial visits.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 to 40 years of age, inclusive
* Judged to be in good health based on medical history, physical examination, vital signs and laboratory tests
* Body mass index (weight kg/m2) between 18 and 35 kg/m2 (inclusive), and body weight between 50 kg and 120 kg (inclusive).
* Willing/able to donate blood (and meets the site's blood donor criteria).
* No severe or significant medical condition and without intercurrent illness (e.g. viral cold or flu, chest infection)
* Not taking any regular oral or intravenous medication.
* Must be willing to abstain from food and caffeine-containing beverages for at least 12 hours beforehand, and alcohol for 24 hours beforehand.

Exclusion Criteria:

* Smoked tobacco or related products within 1 year prior to the study
* Asthmatic
* Occupation with high exposure to air pollution or other inhaled irritant
* Severe or significant medical condition
* Intercurrent illness (e.g. viral cold or flu, chest infection)
* Use of any regular oral or intravenous prescription medication, or non-prescription (including aspirin, ibuprofen, paracetamol, vitamins and herbal supplements), and not at all in the 7 days prior to the study
* Allergy or contraindication to vasodilator drugs (e.g. acetylcholine or sodium nitroprusside)
* Major or traumatic surgery within 12 weeks of screening
* Pregnant or still lactating prior to dose administration (women only)
* Given blood in the 3 months prior to the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Blood eicosanoid levels | Results available within 6 months of final study visit
  Eicosanoids in blood (pg/mL)
Urine eicosanoid levels | Results available within 6 months of final study visit
  Eicosanoids in urine (pg/mL)

SECONDARY OUTCOMES:
blood pressure | Results available immediately at time of measurement
  systolic/diastolic blood pressure (mmHg/mmHg)
Heart rate | Results available immediately at time of measurement
  Heart rate (bpm)
Lung function (FEV1) | Results available immediately at time of measurement
  Forced expiratory volume (% predicted litres)
Lung function (FVC) | Results available immediately at time of measurement
  Forced vital capacity (% predicted litres)
Full blood count | Results available within 3 months of study visit
  Blood cell counts (cells/mL)
Coagulation screen | Results available within 3 months of study visit
  Activated partial thromboplasmin time (seconds)
Internal normailised ratio | Results available within 3 months of study visit
  blood INR (ratio, arbitrary units)
C-reactive protein | Results available within 3 months of study visit
  Serum CRP levels (pg/mL)
Tumour necrosis factor | Results available within 6 months of study visit
  Blood TNFa levels (pg/mL)
Interleukin-6 | Results available within 6 months of study visit
  Blood IL-6 levels (pg/mL)
Blood coagulability (low-shear) | Results available within 6 months of study visit
  Area of thrombus on arterial strip from low sheer-stress Badimon chamber (micrometers squared)
Blood coagulability (high-shear) | Results available within 6 months of study visit
  Area of thrombus on arterial strip from high sheer-stress Badimon chambers (micrometers squared)
Vascular responsiveness (endothelium-dependent vasodilator) | Results available within 1 year of study visit
  Forearm blood flow to acetylcholine (mL blood/mL 100g tissue per min)
Vascular responsiveness (endothelium-independent vasodilator) | Results available within 1 year of study visit
  Forearm blood flow to sodium nitroprusside (mL blood/mL 100g tissue per min)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrews JPM, Joshi SS, Tzolos E, Syed MB, Cuthbert H, Crica LE, Lozano N, Okwelogu E, Raftis JB, Bruce L, Poland CA, Duffin R, Fokkens PHB, Boere AJF, Leseman DLAC, Megson IL, Whitfield PD, Ziegler K, Tammireddy S, Hadjidemetriou M, Bussy C, Cassee FR, Newby DE, Kostarelos K, Miller MR. First-in-human controlled inhalation of thin graphene oxide nanosheets to study acute cardiorespiratory responses. Nat Nanotechnol. 2024 May;19(5):705-714. doi: 10.1038/s41565-023-01572-3. Epub 2024 Feb 16. PMID 38366225